CLINICAL TRIAL: NCT02427191
Title: A Prospective, Single-Blinded, Randomized Controlled Trial of the Micronized dHACM Injection as Compared to the Saline Placebo Injection in the Treatment of Plantar Fasciitis
Brief Title: Micronized dHACM Injectable for the Treatment of Plantar Fasciitis
Acronym: dHACM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIPF004
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Fasciitis, Plantar
Keywords: Chronic plantar fasciitis; Heel pain
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AmnioFix® Injectable (Experimental): 1 mL injection of 40 mg Micronized dehydrated human amnion/chorion membrane (dHACM)
  Interventions: Other: AmnioFix® Injectable
- Saline Injection (Placebo Comparator): Injection of 1mL 0.9% Sodium Chloride Injection, USP
  Interventions: Drug: Saline Injection

INTERVENTIONS:
Other: AmnioFix® Injectable — 1 mL injection of 40 mg Micronized dehydrated human amnion/chorion membrane (dHACM)
  Other Names: dHACM
  Arms: AmnioFix® Injectable
Drug: Saline Injection — Injection of 1mL 0.9% Sodium Chloride Injection, USP
  Other Names: 0.9% NaCl; Normal Saline
  Arms: Saline Injection

SUMMARY:
Prospective, single-blinded, randomized controlled trial of the micronized dHACM injection as compared to the saline placebo injection in the treatment of plantar fasciitis

DETAILED DESCRIPTION:
Approximately 146 patients will be enrolled in this study. Each patient will receive 1 injection and be evaluated for efficacy and safety during a 12-month observation period. The study is expected to be completed within 36 months, inclusive of enrollment and follow-up of all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of plantar fasciitis for ≥ 1 month (30 days) and ≤ 18 months by the investigator
2. VAS Pain scale of ≥ 45 mm at randomization
3. Plantar fasciitis with conservative treatment for ≥ 1 month (30 days), including any of the following modalities:

   * RICE
   * Stretching exercises
   * NSAIDs
   * Orthotics
4. Diagnostic X-Ray within 6 months of enrollment showing view of calcaneus negative for calcaneal fracture or structural abnormalities
5. BMI ≤ 40 kg/m2
6. Age ≥ 21 years and < 80
7. Ability to sign Informed Consent and Release of Medical Information Forms

Exclusion Criteria:

1. Prior surgery or trauma to the affected site
2. Subjects requiring bilateral plantar fasciitis treatment at time of enrollment
3. Prior use of any lower limb injection therapy, including corticosteroids or PRP in either limb within the last 3 months
4. Has diabetes either Type I or Type II
5. Systemic disorders associated with enthesopathy (disorder of entheses, i.e. bone attachments) such as Gout, Reiter's syndrome, rheumatoid arthritis, etc.
6. The presence of comorbidities that can be confused with or can exacerbate the condition- to be assessed by X-ray - including but not limited to:

   * Calcaneal stress fracture
   * Nerve entrapment syndrome (Baxter Nerve Syndrome)
   * Fat pad atrophy
   * Acute traumatic rupture of the plantar fascia
   * Calcaneal tumor
   * Tarsal tunnel syndrome
   * Significant bone deformity of the foot that may interfere with the study
7. Affected site exhibits clinical signs and symptoms of infection
8. Known allergy or known sensitivity to Aminoglycosides, such as Gentamicin sulfate or Streptomycin sulfate
9. Clinically significant abnormal laboratory tests at baseline, including CBC, PT/PTT/INR, liver function and creatinine, as determined by the investigator
10. Patients who are non-ambulatory
11. History of more than 14 days treatment with immuno-suppressants (including systemic corticosteroids) or cytotoxic chemotherapy within 30 days prior to enrollment, or who are anticipated to require such medications during the course of the study
12. Prior radiation at the site
13. Use of any investigational drug(s) or therapeutic device(s) within 3 months preceding enrollment
14. Immune disorders including Systemic Lupus Erythematosus (SLE), Fibromyalgia, Acquired Immunodeficiency Syndrome (AIDS) or Human Immunodeficiency Virus (HIV)
15. History of any condition (including drug or alcohol abuse, medical or psychiatric condition) that is likely to impair understanding of or compliance with the study protocol, in the judgment of the investigator
16. Pregnancy at enrollment or within last 6 months, women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence)
17. Workers' compensation patients

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
20% improvement over baseline Visual Analog Scale for Pain | 3 Months
  Visual Analog Scale
Incidence of adverse events | 12 months
  Review AE at every visit

SECONDARY OUTCOMES:
20% improvement in Foot Function Index-Revised (FFI-R) score from baseline | 3 months
  Foot Function Index
Blood sample analysis for immuno-compatibility of first 20 patients in each treatment arm | 3 and 12 months
  Lab blood draws
Long-term FFI-R outcomes | 6 and 12 months
  Foot Function Index
Long-term Visual Analog Scale (VAS) Pain outcomes | 6 and 12 months
  Visual Analog Scale
Long-term blood sample analysis for immuno-compatibility of first 20 patients in each treatment arm | 6 and 12 months
  Lab blood draws

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Miller, MD, Principal Investigator — MedStar Union Memorial Hospital, Baltimore, MD
Locations (11):
- United States (11):
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Limb Preservation Platform, Inc., Fresno, California
  - Center for Clinical Research, Inc., San Francisco, California
  - Orlando VA Healthcare System, Orlando, Florida
  - Edward Hines Jr. Veterans Administration Hospital, Chicago, Illinois
  - James A. Lovell Federal Health Care Center, North Chicago, Illinois
  - Timonium Foot and Ankle Center, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - WJB Dorn VA Medical Center, Columbia, South Carolina
  - Scott & White Healthcare, Temple, Texas
  - Coastal Podiatry Group, Virginia Beach, Virginia